CLINICAL TRIAL: NCT01791296
Title: The Effect of a Dexmedetomidine-focussed Sleep Protocol* on Delirium Incidence and Healthcare Costs in Critically Ill Patients: A Prospective Randomized, Double-blind, Pilot Study.
Brief Title: Does Nightly Dexmedetomidine Improve Sleep and Reduce Delirium in ICU Patients?
Acronym: SKY-DEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Tufts Medical Center (Other); Northeastern University (Other)
Responsible Party: Principal Investigator, Yoanna Skrobik, Yoanna Skrobik MD FRCP(c), Professor of Medicine, University of Montreal; Lise and Jean Saine critical care chair, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10053
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Sleep Deprivation; Delirium
Keywords: sedation; sleep; delirium; critical illness; sub-syndromal delirium; intensive care
MeSH Terms: conditions — Sleep Deprivation; Delirium; Critical Illness | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding for participants, care providers, investigator and outcomes assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine 0.2-0.7 mcg/kg/hr from 21:30 to 6:00
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Normal Saline 0.2-0.7 mcg/kg/hr from 21:30 to 6:00
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — At 21:30h, all current IV sedatives (whether continuous or intermittent) will be decreased by 50% and study drug started at 0.2 mcg/kg/hour at 21h30 to allow sleep between 22h00 and 6h00. Study infusion will be halved at 6:00am and d/c at 6:15am. The infusion rate will be increased by 0.1mcg/kg/hour every 15 minutes when the Riker-SAS is ≥ 4 up to a maximum rate of 0.7 mcg/kg/hr until the targeted sedation goal of a Riker-SAS of 3 is reached. For agitation (ie., Riker-SAS ≥ 5), 'as needed' IV midazolam (1-5 mg IV q1h prn agitation) may be administered during the upwards titration of the study medication. Administration of any dose of as needed IV midazolam will result in the increase of the study medication by 0.1 mcg/kg/hr when ≥ 15 minutes have elapsed since the last upwards titration.
  Other Names: Precedex
  Arms: Dexmedetomidine
Other: Placebo — At 21:30h, all current IV sedatives (whether continuous or intermittent) will be decreased by 50% and study drug started at 0.2 mcg/kg/hour at 21h30 to allow sleep between 22h00 and 6h00. Study infusion will be halved at 6:00am and d/c at 6:15am. The infusion rate will be increased by 0.1mcg/kg/hour every 15 minutes when the Riker-SAS is ≥ 4 up to a maximum rate of 0.7 mcg/kg/hr until the targeted sedation goal of a Riker-SAS of 3 is reached. For agitation (ie., Riker-SAS ≥ 5), 'as needed' IV midazolam (1-5 mg IV q1h prn agitation) may be administered during the upwards titration of the study medication. Administration of any dose of as needed IV midazolam will result in the increase of the study medication by 0.1 mcg/kg/hr when ≥ 15 minutes have elapsed since the last upwards titration.
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
Specific Aims

1. Establish the feasibility of larger trial by implementing a sleep protocol in the ICU at 2 different sites. Specifically will be estimating the recruitment rates of patients and the compliance with both interventions.
2. Measure the safety and tolerance of adding night-time sedation with dexmedetomidine using adverse effects and withdrawal rates as indicators.
3. Measure the effect of nocturnal dexmedetomidine on pertinent clinical outcomes and use this outcome data to plan a larger, multicenter trial in this area.

The goal of this study is to determine whether a night-time protocol that incorporates a pharmacologic intervention associated with improved sleep (i.e. dexmedetomidine) will improve sleep quality and reduce the incidence of delirium and sub-syndromal delirium in critically ill patients.

DETAILED DESCRIPTION:
The goal of this study is to determine whether a nocturnal protocol that incorporates a pharmacologic intervention associated with improved sleep (i.e. dexmedetomidine) will improve sleep quality and reduce the incidence of delirium and sub-syndromal delirium in critically ill patients where ventilator settings have been optimized to optimize sleep quality.

1. To evaluate the impact of a dexmedetomidine-focussed nocturnal sleep protocol that minimizes arousal from sleep on:

   1. incidence of delirium [Intensive Care Delirium Screening Checklist (ICDSC) score ≥ 4]
   2. incidence of sub-syndromal delirium (ICDSC score 1-3)
   3. outcomes specifically defined by place of discharge from hospital (i.e., home,rehabilitation, or long-term care)
2. To gain an understanding of the effect of night-time sedation with dexmedetomidine on:

   1. patient safety
   2. self-reported sleep quality
   3. sleep quality and architecture [based on a subgroup of 10 patients at Tufts Medical Center who will be evaluated using polysomnography(PSG) for one night]
   4. time spent within targeted sedation goal
   5. time spent without pain
   6. agitation-related events
   7. length of stay in the ICU
   8. duration of mechanical ventilation
   9. length of hospital stay
   10. total health care costs by measuring medication costs and hospitalization costs, as well as calculating effectiveness (sleep, sedation and pain management vs. cost).

This multicenter study will be performed at:

1. Hopital Maissonneuve Rosemont, Montreal, PQ
2. Tufts Medical Center, Boston, MA

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Current expectation on the part of the patient's admitting intensivist for patients to require ICU care for >/= 48 hrs
3. Administered at least one sedative dose (scheduled or prn).

Exclusion Criteria:

1. Patients with delirium (intensive care delirium screening checklist score ≥ 4) or disorientation (not oriented to person and/or place)
2. Patients in whom an ICDSC cannot be reliably completed (e.g. primary language is not French or English, baseline severe hearing impairment)
3. Inability by one of the investigators to obtain informed consent from the legally authorized representative
4. Treating physician refusal
5. Heart rate ≤ 50 BPM
6. Systolic blood pressure ≤ 90 mmHg despite the administration of norepinephrine ≥ 15 mcg/min and/or vasopressin ≥ 0.04 units/min
7. Admission with acute decompensated heart failure
8. History of heart block without pacemaker based on hospital admission note.
9. Acute alcohol withdrawal based on hospital admission note
10. History of end stage liver failure (based on presence of ≥ 1 or more of the following: AST/ALT ≥ 2 times ULN, INR ≥ 2, total bilirubin ≥ 1.5)
11. Irreversible brain disease consistent with severe dementia based on hospital admission note
12. Pregnancy (all women of child-bearing age will undergo a pregnancy test prior to study enrolment)
13. Known allergy or sensitivity to clonidine or dexmedetomidine
14. Current treatment with dexmedetomidine

p. Prognosis considered to be hopeless based on consultation with the ICU admitting physician q. Age ≥80 years r. Currently being managed with a high frequency oscillating mode (HFOV) of mechanical ventilation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Development of delirium | participants will be followed for the duration of their ICU stay, an expected average of 5-7 days
  Delirium will be assessed with the ICDSC (Intensive Care Delirium Screening CHecklist) q12h [Delirium = ICDSC score >/= 4]

SECONDARY OUTCOMES:
Development of subsyndromal delirium | participants will be followed for the duration of ICU stay, an expected average of 5-7 days
  ICDSC measurement (routine in all participating units) q12h [Subsyndromal delirium = ICDSC of 1-3]

OTHER OUTCOMES:
Sleep quality | participants will be followed for the duration of ICU stay, an expected average of 5-7 days
  Sleep quality will be assessed with a validated sleep questionnaire and polysomnography (PSG) evaluation in a subset of 10 patients at Tufts Med Center site

CONTACTS AND LOCATIONS:
Overall Officials: Yoanna Skrobik, MD, Principal Investigator — Université de Montréal
Locations (2):
- Tufts Medical Center, Boston, Massachusetts, United States
- Maisonneuve Rosemont Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Duprey MS, Devlin JW, Skrobik Y. Is there an association between subjective sleep quality and daily delirium occurrence in critically ill adults? A post hoc analysis of a randomised controlled trial. BMJ Open Respir Res. 2020 Aug;7(1):e000576. doi: 10.1136/bmjresp-2020-000576. PMID 32847946
- [Derived] Skrobik Y, Duprey MS, Hill NS, Devlin JW. Low-Dose Nocturnal Dexmedetomidine Prevents ICU Delirium. A Randomized, Placebo-controlled Trial. Am J Respir Crit Care Med. 2018 May 1;197(9):1147-1156. doi: 10.1164/rccm.201710-1995OC. PMID 29498534